CLINICAL TRIAL: NCT01769339
Title: Effectiveness and Safety of Daktacort Feminine Care Cream in the Treatment of Vulvar Candidiasis
Brief Title: An Efficacy and Safety Study of Miconazole and Hydrocortisone Cream in the Treatment of Vulvar Candidiasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015721; MICFUN4001
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Results first posted 2013-03-25 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-02

CONDITIONS: Vulva; Candidiasis
Keywords: Vulvar Candidiasis; Miconazole; Hydrocortisone; Daktacort Feminine Care Cream
MeSH Terms: conditions — Candidiasis | interventions — Miconazole; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Miconazole plus Hydrocortisone (Experimental)
  Interventions: Drug: Miconazole plus Hydrocortisone

INTERVENTIONS:
Drug: Miconazole plus Hydrocortisone — Participants will apply miconazole plus hydrocortisone cream topically to the lesion twice daily up to Day 14 by rubbing gently until it has been completely penetrated into the affected vulvar (the tissues around the opening to the vagina) area and the treatment should be continued without interruption. Participants will be assessed for signs and symptoms of vulvar candidiasis at Day 14. Medication will be continued till Day 28, if signs and symptoms of vulvar candidiasis are not cured clinically on Day 14.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of miconazole plus hydrocortisone cream in the treatment of participants with vulvar candidiasis (yeast infection of the vulva).

DETAILED DESCRIPTION:
This is an open label (all people know the identity of the intervention), single-arm, prospective (study following participants forward in time) study to evaluate the efficacy and safety of miconazole plus hydrocortisone cream in participants with vulvar candidiasis. Participants will be evaluated and assessed on the degree of pruritus (itchiness) and screened for candidiasis on the baseline. Participants will apply the cream once enrolled and will be assessed for 1-hour to get the time to relief. Each participant will apply the study medication topically (applied to skin) to the lesion twice daily up to Day 14 by rubbing gently until it has been completely penetrated into the vulvar area affected and the treatment should be continued without interruption. Participants will be followed-up after 14 days and will be assessed clinically for signs and symptoms of vulvar candidiasis; if not cured, participants will continue the medication up to Day 28. Primary efficacy endpoint will be the time needed to achieve pruritus relief. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria: - Positive potassium hydroxide (KOH) mount / Gram stain (a method used to diagnose bacterial infection) of vulvar (the tissues around the opening to the vagina) scrapings - Vulvar candidiasis with at least mild pruritus Exclusion Criteria: - Participants with vaginal candidiasis (yeast infection of the vagina) - History of allergy to miconazone (an antifungal agent, is used for skin infections such as vaginal yeast infections) and/or other components of the study drug - Pruritus caused by etiologic (the cause) agents aside from fungi - Tuberculous (bacterial infection that usually results in a serious lung disorder) skin infection - Herpes simplex (viral infection), vaccinia (vaccine used to eradicate smallpox), all forms of varicella (infection caused by the varicella-zoster virus), and vulvar malignancy (cancer)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica Clinical Trial, Study Director — Janssen Pharmaceutica

RESULTS

PARTICIPANT FLOW:
Groups:
- Miconazole Plus Hydrocortisone: Participants applied miconazole plus hydrocortisone cream topically (applied to skin) to the lesion twice daily up to Day 14. Treatment continued till Day 28, if signs and symptoms of vulvar candidiasis (yeast infection of the vulva) were not cured clinically on Day 14.
Period: Overall Study
Arm/Group | Miconazole Plus Hydrocortisone
Started | 115
Completed | 72
Not Completed | 43
Not completed — Lost to Follow-up | 42
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Miconazole Plus Hydrocortisone: Participants applied miconazole plus hydrocortisone cream topically to the lesion twice daily up to Day 14. Treatment continued till Day 28, if signs and symptoms of vulvar candidiasis were not cured clinically on Day 14.
Arm/Group | Miconazole Plus Hydrocortisone
Number analyzed (Participants) | 115
Age Continuous [Mean (Standard Deviation); unit: years] | 37.76 (9.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Time to Itch Relief
Description: Time to itch relief is defined as time needed to achieve pruritus (itchiness) relief.
Time Frame: 1-hour after initial application
Population: Analysis population included all the participants who received at least 1 dose of study medication.
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Miconazole Plus Hydrocortisone
Number analyzed (Participants) | 115
minutes | 13.36 (1.41)

2. Secondary Outcome: Percentage of Participants Who Achieved Clinical Cure
Description: Participants were considered as clinically cured if the potassium hydroxide (KOH) mount / Gram stain (a method used to diagnose bacterial infection) test was negative for infection.
Time Frame: Baseline up to Day 28
Population: Analysis population included all the participants who received at least 1 dose of study medication. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Miconazole Plus Hydrocortisone
Number analyzed (Participants) | 74
percentage of participants | 97.30

3. Secondary Outcome: Modified Itch Severity Scale (MISS) Score
Description: The MISS is a specific instrument for assessing and quantifying the intensity of pruritus. The MISS score ranges from 0 to 21, where 0=no itching and 21=very severe itching.
Time Frame: Baseline and Day 28
Population: Analysis Population included all the participants who received at least 1 dose of study medication. Here 'n' signifies those participants who were evaluable at specified time-point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Miconazole Plus Hydrocortisone
Number analyzed (Participants) | 115
units on a scale
  Baseline (n=115) | 7.25 (2.57)
  Day 28 (n=7) | 4.27 (0.63)
Statistical Analysis 1: Comparison: Miconazole Plus Hydrocortisone; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

4. Secondary Outcome: Pruritus Symptom Assessment by Visual Analog Scale (VAS) Score
Description: Pruritus is assessed by using a 100 millimeter (mm) of VAS score ranges from 0 to 100 mm, where 0 mm=no pruritus and 100 mm=worse pruritus.
Time Frame: 1-hour after initial application
Population: Data was not collected as only few participants had pruritus after 1-hour of study drug application.
Arm/Group | Miconazole Plus Hydrocortisone
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From signing of informed consent until 30 days after the last dose of study medication
Arm/Group | Miconazole Plus Hydrocortisone
Serious Adverse Events (participants affected / at risk) | 0/115
Other Adverse Events (participants affected / at risk) | 2/115
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Miconazole Plus Hydrocortisone (N=115)
Pruritus (Skin and subcutaneous tissue disorders) | 2

LIMITATIONS AND CAVEATS:
Data was not collected for pruritus symptom assessment by visual analog scale outcome measure as only few participants had pruritus after 1-hour of study drug application.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No